CLINICAL TRIAL: NCT03175172
Title: A Phase 2 Single-arm Study to Evaluate Safety and Efficacy of CRS-207 With Pembrolizumab in Adults With Previously-Treated Malignant Pleural Mesothelioma
Brief Title: Evaluation of CRS-207 With Pembrolizumab in Previously Treated Malignant Pleural Mesothelioma (MPM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to low enrollment and lack of clinical activity.
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-13; KEYNOTE KN-701 (Other: (Other Identifier: Merck Sharp & Dohme Corp))
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2019-02-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): CRS-207 and pembrolizumab will be administered in 3-week cycles. For Cycle 1, pembrolizumab (200 mg) will be administered by intravenous (IV) infusion over 30 minutes on Day 1 and CRS-207 (starting dose 1 × 10e9 colony-forming units [CFU]) will be administered by IV infusion over 1 hour on Day 2. If the infusions are well tolerated, pembrolizumab and CRS-207 may be administered on the same day (Day 1) for subsequent cycles. After 4 cycles, pembrolizumab will continue to be administered on Day 1 at each treatment cycle (every 3 weeks); CRS-207 will be administered once every 6 weeks (every other cycle). Treatment will continue for up to 35 cycles as long as there is adequate safety and potential for clinical benefit.
  Interventions: Biological: CRS-207; Biological: Pembrolizumab

INTERVENTIONS:
Biological: CRS-207 — Administered by IV infusion over approximately 1 hour.
Biological: Pembrolizumab — Administered by IV infusion over approximately 30 minutes.
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to evaluate whether CRS-207 with pembrolizumab is safe and effective in adults with MPM who have failed prior anti-cancer therapy.

DETAILED DESCRIPTION:
The population for this study will consist of approximately 35 adults with histologically-confirmed MPM (epithelial or biphasic) whose disease has progressed after 1-2 prior anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed epithelial or biphasic MPM; biphasic tumors must have a predominantly (≥50%) epithelial component
2. No more than 2 prior lines of anti-cancer therapy, one of which must have included pemetrexed and a platinum.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
4. Adequate organ and marrow function
5. Adequate lung function; forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) ≥ 45% of predicted value as measured by spirometry; and oxygen saturation ≥ 90% on room air

Exclusion Criteria

1. Pleurodesis within 14 days prior to first dose of study drug
2. Receiving tumor necrosis factor (TNF) pathway inhibitors, PI3 kinase inhibitors, systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
3. Active secondary malignancy
4. Prior anti-cancer monoclonal antibody within 4 weeks prior to first dose of study drug, or not recovered from adverse effects due to agents administered more than 4 weeks earlier
5. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to first dose of study drug
6. History of (non-infectious) pneumonitis that required steroids or current pneumonitis
7. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent, or agents targeting other checkpoint pathways (e.g. CTLA-4)
8. Prior immunotherapy with CRS-207 or any other Listeria-based agent, therapeutic cancer vaccine, or adoptive T cell immunotherapy
9. Implanted medical devices that pose high risks for colonization and cannot be easily removed (e.g., artificial heart valves, pacemakers, prosthetic joints, orthopedic screw(s), metal plate(s)) if infection occurs. Other common devices such as venous access devices (e.g., Port-a-Cath or Mediport) may be permitted as well as arterial and venous stents and dental and breast implants that were placed more than 3 months prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - NIH National Cancer Institute, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne MJ, Nowak AK. Modified RECIST criteria for assessment of response in malignant pleural mesothelioma. Ann Oncol. 2004 Feb;15(2):257-60. doi: 10.1093/annonc/mdh059. PMID 14760119

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: CRS-207 and pembrolizumab were administered in 3-week cycles. For Cycle 1, pembrolizumab (200 mg) was administered by intravenous (IV) infusion over 30 minutes on Day 1 and CRS-207 (starting dose 1 × 10e9 colony forming units [CFU]) was administered by IV infusion over 1 hour on Day 2. If tolerated, pembrolizumab and CRS-207 were administered on the same day (Day 1) for subsequent cycles. After 4 cycles, pembrolizumab continued to be administered on Day 1 at each treatment cycle (every 3 weeks); and CRS-207 was administered once every 6 weeks (every other cycle).
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 0
Not Completed | 10
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated by Sponsor | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis provided for all subjects who were administered at least 1 dose of protocol-specified drug (the Safety Analysis Set [SAF]).
Groups:
- Experimental: CRS-207 and pembrolizumab were administered in 3-week cycles. For Cycle 1, pembrolizumab (200 mg) was administered by IV infusion over 30 minutes on Day 1 and CRS-207 (starting dose 1 × 10e9 CFU) was administered by IV infusion over 1 hour on Day 2. If tolerated, pembrolizumab and CRS-207 were administered on the same day (Day 1) for subsequent cycles. After 4 cycles, pembrolizumab continued to be administered on Day 1 at each treatment cycle (every 3 weeks); and CRS-207 was administered once every 6 weeks (every other cycle).
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 7
  Other | 1
  Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was evaluated based upon the best overall response (BOR) for individual study subjects. BOR was determined by the highest post-baseline qualitative response value for each assessed subject as measured by modified response evaluation criteria in solid tumors (modified RECIST) for MPM (Byrne and Nowak, 2004) and given the following hierarchy of overall response results: complete response (CR) > partial response (PR) > stable disease (SD) > progressive disease (PD) > not evaluable (NE). The protocol-specified ORR was defined as the percentage of evaluable subjects with a BOR of CR or PR; however, this percentage was not calculated per the final study Statistical Analysis Plan (SAP). Therefore, the number of evaluable subjects with BOR RECIST v1.1 values of CR, PR, SD, PD, and NE are provided for this outcome measure.
Time Frame: BOR was assessed from the first dose of study treatment until documented disease progression, initiation of new cancer treatment, death, or study termination, whichever is earlier, assessed up to 15 weeks.
Population: Analysis based on subjects who received ≥1 dose of study treatment and had ≥1 evaluable post-baseline modified RECIST for MPM tumor response assessment or were discontinued due to toxicity (the Evaluable Analysis Set [EAS]). 1 subject did not have post-baseline tumor response assessments and could not be evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 8
  Not Evaluable | 0

2. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of evaluable subjects who exhibited a post-baseline tumor assessment BOR rating of CR, PR, or SD per modified RECIST for MPM.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 6
  Not Evaluable | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Number of weeks from the date of first dose of study treatment to the first date of objectively determined progressive disease (PD) (per modified RECIST for MPM) or death from any cause, estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CI). Subjects who do not experience PD and are alive on or before the data cut-off date will be censored at the time of last tumor assessment or data cut-off date, whichever is earlier.
Time Frame: Subjects followed for disease progression from first dose of study treatment until documented disease progression, initiation of new cancer treatment, death, or study termination, whichever is earlier, assessed up to 9 weeks.
Population: Analysis of PFS was performed on subjects in the SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Experimental
Number analyzed (Participants) | 10
weeks | 6 [3.43 to 7.14]

4. Secondary Outcome: Improvement in Pulmonary Function
Description: Percentage of subjects with improvement in forced vital capacity (FVC), defined as an increase from baseline of either ≥400 mL or ≥20% assessed using spirometry
Time Frame: Subjects tested by spirometry at Screening and up to 7 days prior to dosing every other cycle starting at Cycle 3 until 4 weeks post final dose, assessed up to 16 weeks.
Population: Analysis of FVC was performed on all subjects in the SAF. No subjects showed improvement in FVC.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Number of weeks from the date of first dose of study treatment to the date of death from any cause, estimated using KM methods with 95% CIs for subjects in the SAF. Subjects without documentation of death at the time of analysis were censored as of the date the subject was last known to be alive, or the data cut-off date, whichever is earlier.
Time Frame: OS was assessed from the first dose of study treatment until death or study termination, whichever is earlier, assessed up to 25 weeks.
Population: Analysis of OS was performed on subjects in the SAF.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Experimental
Number analyzed (Participants) | 10
weeks | 12.57 [8.14 to 18.14]

ADVERSE EVENTS:
Time Frame: Subjects were followed for serious and non-serious adverse events (AEs) from the beginning of any study drug until 28 days following the last dose of study drug or initiation of a subsequent cancer-related therapy, whichever is earlier, an average of 3 months. Subjects were followed for survival for 12 months after end-of-treatment (EOT) or until study termination on 31 January 2018, whichever is earlier, an average of 14 weeks.
Description: AEs reported for the SAF. Methods of determining whether certain AEs have occurred include regular investigator assessment and regular laboratory testing.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=10)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
HYPOTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=10)
CHILLS (General disorders) | 10
PYREXIA (General disorders) | 9
OEDEMA PERIPHERAL (General disorders) | 3
FATIGUE (General disorders) | 2
OEDEMA (General disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DRY MOUTH (Gastrointestinal disorders) | 1
HYPOTENSION (Vascular disorders) | 4
HOT FLUSH (Vascular disorders) | 1
HYPERTENSION (Vascular disorders) | 1
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 2
BLOOD CREATININE INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
TACHYCARDIA (Cardiac disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1
CANDIDA INFECTION (Infections and infestations) | 1
GINGIVITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
DYSGEUSIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
RESTLESSNESS (Psychiatric disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1
BREAST OEDEMA (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated early and included a small number of subjects, and insufficient data were available to evaluate the clinical activity of the study treatment. Due to low enrollment, some protocol-specified outcome measures were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction is that study results will first be published in a joint multi-center paper unless (a) written confirmation is provided to the site or PI indicating that there will be no multi-center publication, or (b) at least 15 months have passed after the completion of data analysis at all study sites. Publications will be submitted for sponsor review ≥ 30 days prior to the publication date. Sponsor cannot require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03175172/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT03175172/SAP_001.pdf